CLINICAL TRIAL: NCT06944262
Title: Évaluation de la détresse Post-traumatique Relative au Cancer Dans l'année Suivant le Diagnostic Chez Les Patients et Les Aidants et Identification de Leurs Attentes Envers un Accompagnement personnalisé
Brief Title: Assessment of Cancer-related Post-traumatic Stress in Patients and Caregivers in the Year Following Diagnosis, and Identification of Their Expectations of Personalized Support - CANDYSTRESS
Acronym: CANDYSTRESS
Status: Recruiting | Type: Observational
Sponsor: Lille University (Other)
Collaborators: Centre Oscar Lambret, Lille, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: D2023-02
Record Dates: First submitted 2025-04-03; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Healthcare Professionnals; Caregiver Distress; Caregiver; Caregiver Stress Syndrome
Keywords: cancer; trauma; patients; caregivers; dyad; cancer-related post-traumatic stress disorder
MeSH Terms: conditions — Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Part 1 - patients groups: (n = 150) = Male or female, 18 years of age or older, recently (<4 months) diagnosed with breast, gynecological, testicular or digestive cancer at the time of the announcement visit (i.e., the announcement to the patient of the treatment plan after the initial multidisciplinary consultation meeting in the cancer center)
- Part 1 - caregivers group: (n = 150) = Men or women aged 18 or over, designated by the patient as their primary caregiver (i.e. "a family member, friend or other person who has helped care for you since your diagnosis")
- Part 2 - patients: Men or women of legal age who have or have had cancer, Members of a local patient association or of the Oscar Lambret Center's "patient partners" committee.
  For each type of participant (patients, caregivers, healthcare professionals), 3 focus groups will be set up to collect a sufficient amount of data to reach data saturation (Guest et al., 2017; Wilkinson, 2013). In all, 9 focus groups will be set up. Each group will have between 4 and 8 participants.
- Part 2 - caregivers: Men or women of legal age who are or have been caregivers for a cancer patient, members of a local caregivers' association.
  For each type of participant (patients, caregivers, healthcare professionals), 3 focus groups will be set up to collect a sufficient amount of data to reach data saturation (Guest et al., 2017; Wilkinson, 2013). In all, 9 focus groups will be set up. Each group will have between 4 and 8 participants.
- Part 2 - healthcare professionals: Medical and paramedical staff at the Oscar Lambret Center Or non-hospital personnel involved in the medical or psychological care of patients, Professionals not involved in the present study.
  For each type of participant (patients, caregivers, healthcare professionals), 3 focus groups will be set up to collect a sufficient amount of data to reach data saturation (Guest et al., 2017; Wilkinson, 2013). In all, 9 focus groups will be set up. Each group will have between 4 and 8 participants.

SUMMARY:
The impact of cancer on the lives of patients and their caregivers is undeniable. In addition to the potentially traumatic aspects (i.e., creating a very violent emotional shock) linked to the announcement of the disease and the various stages of the care pathway (effects of treatment, announcement of a cancer recurrence), even before the onset of the disease, patients and their caregivers may have been directly or indirectly confronted with traumatogenic events (e.g., childhood abuse, sudden death). They may therefore be more likely to develop a stress-related mental disorder in their lifetime. The question of the accumulation of traumatic events, the identification of groups of people at risk of developing symptoms of distress, and the management of these symptoms is therefore crucial. In addition, the mutual influence within the patient-caregiver dyad in terms of emotional adjustment, and its evolution throughout the cancer care pathway, are key elements to be considered in these issues.

The CandyStress project is based on a partnership with patients, their caregivers and carers to identify the needs of patient-caregiver dyads at risk of cancer-related post-traumatic stress disorder (Ca-PTS). Longitudinal screening for Ca-PTS in the year following cancer diagnosis will be carried out to identify the characteristics of at-risk dyads who could benefit from long-term support. The aim of this project is to identify the potential need for targeted support and the desired format of this support. This is a preliminary step in identifying needs and the context conducive to the implementation of personalized support, but in no way an evaluation of the effectiveness of an intervention.

ELIGIBILITY:
Inclusion Criteria:

Part 1. Diagnosis of Ca-PTS

Patient inclusion criteria:

* Male or female, 18 years of age or older,
* recently (<4 months) diagnosed with breast, gynecological, testicular or digestive cancer at the time of the announcement visit (i.e., the announcement to the patient of the treatment plan after the initial multidisciplinary consultation meeting in the cancer center - in accordance with the Cancer Plan),
* with cancer requiring oncological treatment,
* starting oncology treatment at the Oscar Lambret Center,
* with no Central Nervous System (CNS) metastases,
* with a PRONOPALL score ≤3 (favorable prognosis group, Bourgeois et al., 2017) or expected survival greater than 6 months,
* who have given signed consent to participate in the study and are covered by French social security,
* able to identify a caregiver (i.e., a family member, friend or other person who has helped care for them since diagnosis).
* equipped with a computer or tablet equipped with a webcam and an internet connection, for the online questionnaire - the webcam is only necessary if the participant wants the IGE to be present via video on the computer, if they prefer the video to be made over the phone, in which case they must also be equipped with a smartphone enabling video calls.

Inclusion criteria for caregivers:

* Male or female, 18 years of age or older,
* designated by the patient as their primary caregiver (i.e. "a family member, friend or other person who has helped care for you since diagnosis"),
* have given their signed consent to participate in the study.
* equipped with a computer or tablet equipped with a webcam and an internet connection, for the online questionnaire - the webcam is only necessary if the participant wishes the IGE to be present via video on the computer, if he/she prefers the video to be made over the phone, in which case it is also necessary to be equipped with a smartphone enabling video calls.

Part 2. Gathering expectations for personalized support and its components.

In addition, 3 types of focus groups will be set up remote :

Focus groups with patients from local associations, as well as patient partners of the Oscar Lambret Center and patients from Part 1 if they are interested.

Inclusion criteria for patient focus groups:

* Men or women of legal age who have or have had cancer,
* Members of a local patient association or of the Oscar Lambret Center's "patient partners" committee,
* Or have participated in part 1 (Ca-PTS screening, once the 3 steps have been completed),
* Equipped with a computer or tablet with camera and internet connection,
* Have given their consent to take part in the study.

Focus group with caregivers from local associations as well as "partner caregivers" from the Oscar Lambret Center and caregivers from part 1 if they are interested.

Inclusion criteria for "caregiver" focus groups:

* Men or women of full age who are, or have been, caregivers of a cancer patient,
* members of a local caregivers' association,
* or having participated in part 1 (Ca-PTS screening, once the 3 steps have been completed),
* Equipped with a computer or tablet with camera and internet connection,
* Having given their consent to take part in the study.

Focus groups with hospital medical and paramedical staff as well as non-hospital caregivers involved in the medical in the medical and psychological follow-up of patients.

Inclusion criteria for caregiver focus groups:

* Member of the medical and paramedical staff of the Oscar Lambret Center
* Or non-hospital staff involved in the medical or psychological care of patients,
* Professionals not involved in the present study,
* Equipped with a computer or tablet with camera and internet connection
* Having given their consent to participate in the study

Exclusion Criteria:

Part 1. Diagnosis of Ca-PTS

Non inclusion criteria for patients :

* Patients with meningeal or cerebral metastases,
* Patients with cancer recurrence,
* Patients suffering from a psychiatric or neurological disorder likely to impair their ability to reason or judge (in particular psychotic disorder, autism spectrum disorder, intellectual disability),
* Patients with a psychological or physical incapacity to answer questionnaires, certified by medical staff,
* Patients subject to a custodial sentence, guardianship or protection of vulnerable adults,
* Presence of CNS metastases (risk of cognitive impairment preventing completion of questionnaires).

Non-inclusion criteria for caregivers:

* Caregivers suffering from a psychiatric or neurological disorder likely to impair their ability to reason or exercise judgment judgment (in particular psychotic disorder, autism spectrum disorder intellectual disability), or for whom there is a suspicion (not there is a suspicion (no additional examination is prescribed to confirm this criterion, which remains self-declaratory).
* Caregivers with a psychological or physical inability to answer questionnaires, or for whom there is a suspicion suspicion (no further tests are required to confirm this criterion which remains self-reported).
* Caregivers subject to a custodial sentence, guardianship or protection guardianship or protection of vulnerable adults.

Part 2. Collection of expectations for personalized support and its components.

Non-inclusion criteria for patients and caregivers who participated in the screening part of the Ca-PTS :

- Failure to complete all measurement times (T0, T1, T2)

Non-inclusion criteria for focus groups (patients, caregivers): none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: centre oscar lambret
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL5) | measured in the month following the announcement of the cancer treatment, then 6 months and 12 months later - in patients and their caregiver
  total score (0-80) reflects the severity of Post Traumatic Stress Disorder (PTSD) symptoms. A score threshold > 32 has been validated as reflecting probable PTSD

SECONDARY OUTCOMES:
self reported general physical condition | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  answer to the item "How do you feel physically impaired at the moment?" (likert scale from 0: "not at all" to 10: "absolutely")
perception of the general physical condition in the other dyad member | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  answer to the item:: "To what extent do you think your loved one feels physically diminished at the moment? " (likert scale from 0: "not at all" to 10: "absolutely")
self reported distress | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  answer to the item "To what extent do you feel psychologically distressed at the moment? " ((likert scale from 0: "not at all" to 10: "absolutely")
perception of the distress in the other dyad member | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  answer to the item: "To what extent do you think your loved one feels psychologically distressed at the moment? " (likert scale from 0: "not at all" to 10: "absolutely")
self reported physical pain (only in patients) | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  answer to the item "to what extent are you currently experiencing physical pain?" (likert scale from 0: "not at all" to 10: "absolutely")
exposure to potentially traumatic events | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  self reported Life Event Checklist for DSM-5 (LEC-5). The total score is 0 to 48. The higher the score, the more the participant reports traumatic events.
post traumatic stress disorder (PTSD) | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  PTSD checklist for DSM 5 (PCL-5). The total score (0-80) reflects the severity of the PSTD symptoms, and a cut off of 32 a possible PTSD.
anxiety symptoms | : from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  Generalized Anxiety Disorder (GAD7). The overall score ranges from 0 to 21. Scores of 5, 10 and 15 represent thresholds for mild, moderate and severe anxiety respectively
depressive symptoms | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  Patient Health Questionnaire (PHQ9). The total score ranges from 0 to 27, with a score of 10 or more indicating moderate depression.
social support | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  Social Support Questionnaire SSQ6. Higher SSQ6 scores reflect greater satisfaction with the level of social support.
difficulties in emotion regulation | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  Difficulties in Emotion Regulation Scale Short Form (DERS SF). The higher the score, the greater the difficulty of emotional regulation.
resilience | from baseline (in the month following the announcement of the cancer treatment) to 6 months and 12 months later
  Resilience Resources Scale (RSS). The total score ranges from 12 to 60. Higher scores reflect greater resilience
Questions about potential personalized support | baseline
  Participants will be asked whether they personally feel the need for psychological support to manage their symptoms, and whether they would be willing to engage in such support. If so, they will be asked to specify when they think this support should be offered, and in what form These answers will be collected using open-ended questions.
Socio-demographic factors | at inclusion (i.e in the month following the announcement of the cancer treatment) - for patients and caregivers
  age, gender, marital status, socio-professional category, level of education

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Oscar Lambret, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815